CLINICAL TRIAL: NCT03303924
Title: A Phase I Study to Determine and Compare Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations of Intravenous ETX2514 and Sulbactam Administered to Healthy Adult Subjects
Brief Title: Study to Determine and Compare Plasma and Intrapulmonary Concentrations of ETX2514 and Sulbactam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS2514-2017-0001
Record Dates: First submitted 2017-08-22; First posted 2017-10-06 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Pharmacokinetic; Bronchoalveolar Lavage; Epithelial Lining Fluid; Alveolar Macrophage; Gram-negative bacterium; Acinetobacter baumannii
MeSH Terms: interventions — durlobactam; Sulbactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ETX2514 and sulbactam (Experimental): Healthy male and female subjects, non-smoking, will receive multiple doses of ETX2514 1.0 g and sulbactam 1 g via intravenous (IV) infusion every 6 hours with each dose of medication infused over 3 hours.
  Interventions: Drug: ETX2514 and sulbactam

INTERVENTIONS:
Drug: ETX2514 and sulbactam — Each subject will receive three doses of of ETX2514 1.0 g and sulbactam 1.0 g via intravenous (IV) infusion administered every 6 hours with each drug infused over 3 hours

SUMMARY:
This is a Phase 1, multiple dose, open-label pharmacokinetic study conducted in healthy adult male and female subjects to determine and compare plasma, epithelial lining fluid (ELF) and alveolar macrophage (AM) concentrations of ETX2514 and sulbactam in healthy adult subjects after intravenous infusion of ETX2514 1.0 g given concurrently with intravenous sulbactam 1.0 g, administered every 6 hours with each infused over 3 hours, for 3 consecutive doses

DETAILED DESCRIPTION:
Blood samples for determining plasma concentrations of ETX2514 and sulbactam will be collected within 5 minutes prior to and at 1.0, 2.0, 2.5, 2.95, 3.05, 3.25, 3.5, 4.0, 5.0 and 6.0 hours after start of the third dose (last dose) administered on Day 2.

Each subject will undergo one standardized bronchoscopy with bronchoalveolar lavage (BAL) in the outpatient bronchoscopy suite at 1.0, 2.5, 3.25, 4.0, or 6.0 hours after start of the infusion of the third dose of ETX2514 and sulbactam (6 subjects per timepoint) on Day 2.

Safety will be assessed throughout the study by adverse event monitoring, clinical laboratory tests, ECG, physical examination, and vital sign monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject, between 18 and 55 years of age (both inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2 and weight between 55.0 and 100.0 kg (both inclusive).
3. Be in general good health without clinically significant medical history as judged by the Principal Investigator.
4. Provide voluntary written informed consent prior to any study procedures and is willing and able to comply with the prescribed treatment protocol and evaluations.
5. Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to screening.
6. Clinical laboratory values within the normal limits as defined by the clinical laboratory, unless the Principal or sub-Investigator decides that out-of-range values are not clinically significant.
7. If male, agree to be sexually abstinent or agree to use two approved methods of contraception when engaging in sexual activity from screening until 90 days following the last administration of the study drug, and to not donate sperm during same time period. In the event that the sexual partner is surgically sterile, contraception is not necessary.
8. Female subjects of child bearing potential must agree to practice two highly effective methods of birth control (as determined by the Investigator; one of the methods must be a barrier technique) from Screening until 30 days after the last dose of study drug.
9. Postmenopausal females (defined as 12 months spontaneous amenorrhea) with serum follicle stimulating hormone levels ≥ 40 mlU/mL or females who have undergone one of the following sterilization procedures at least 6 months prior to screening (and is documented):

   1. Bilateral tubal ligation
   2. Hysterectomy
   3. Hysterectomy with unilateral or bilateral oophorectomy
   4. Bilateral oophorectomy.

Exclusion Criteria:

1. History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antimicrobial (e.g., penicillin, cephalosporin, sulbactam or carbapenem)
2. History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
3. Calculated creatinine clearance less than 60 mL/min (Cockcroft-Gault method) at screening or confinement.
4. Positive alcohol breath test or urine drug screen test at screening or confinement.
5. Positive testing for HIV, Hepatitis B or Hepatitis C.
6. History or presence of alcohol or drug abuse within the 2 years prior to screening.
7. Excessive intake of alcohol, defined as an average daily intake of greater than three units, or an average weekly intake of greater than 21 units (one unit is equivalent to 1 can or bottle (12 oz) of beer, or 1 measure (1.5 oz) of spirits, or 1 glass (5 oz) of wine) in the last 6 months prior to screening.
8. History of allergic or other serious adverse reactions to lidocaine or amide anesthetic agents.
9. Clinically significant pulmonary or any other disease that prevents a subject from undergoing bronchoscopy with pulmonary lavage.
10. Spirometry results showing an forced expiratory volume at one second (FEV1) <80% of predicted.
11. Use of probenecid within 30 days before confinement.
12. Use of medication, except for acetaminophen which is allowed up to 3 days before confinement. Multivitamins and vitamin C are allowed up to 7 days before confinement (Day 1). All other medication (including over the counter medication, health supplements, and herbal remedies such as St. John's Wort extract must have been stopped at least 14 days prior to confinement), unless agreed as non-clinically relevant by the Principal Investigator.
13. Engagement in strenuous activity within 96 hours of confinement (Day 1) until discharge.
14. History of seizures, head injury or meningitis (e.g., epilepsy).
15. History of bleeding disorders.
16. History or evidence of difficulty in donating blood.
17. Use of any prescription medication (with the exception of hormonal contraceptives or hormone replacement therapy for females) within 14 days prior to confinement.
18. Blood donation/plasma donation or significant blood loss (i.e., >500 mL) within 60 days prior to screening.
19. Participation in another investigational drug or device study or treated with an investigational drug within 30 days or five half-lives (whichever is longer) prior to screening.
20. Females who are pregnant or lactating.
21. Surgery within the past three months prior to screening determined by the investigator to be clinically relevant.
22. Any acute illness including clinically significant infection within 30 days prior to screening.
23. Subjects who have any of the following abnormalities on laboratory values at screening or prior confinement including:

    1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL.
    2. Absolute neutrophil count <1,200/mm3, platelet count <120,000/mm3.
24. Unwillingness or inability to comply with the study protocol for any other reason.
25. Use of caffeine or xanthine containing products, Seville oranges (sour), grapefruit or grapefruit juice within 48 hours prior to study drug dosing.
26. Any other condition or prior therapy, which, in the opinion of the Principal Investigator, would make the subject unsuitable for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Mean maximum observed drug concentration (Cmax) in blood | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analysis predose and after the 3 dose. The 3rd dose of ETX2514 and sulbactam will be administered on Day 2
Mean Cmax in epithelial lining fluid (ELF) | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  Bronchoalveolar lavage fluid will be collected for ETX2514SUL PK at 1, 2.5, 3.25, 4, or 6 hours.
Mean area under the curve (AUC) 0-6h in blood | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  AUC0-6h defined as the area under the concentration versus time curve from time zero to 6 hours postdose. Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analysis predose and after the 3 dose. The 3rd dose of ETX2514 and sulbactam will be administered on Day 2
Mean terminal half-life (t1/2) in blood | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analysis predose and after the 3 dose. The 3rd dose of ETX2514 and sulbactam will be administered on Day 2
Mean volume of distribution in the terminal elimination phase (Vdss) in blood | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analysis predose and after the 3 dose. The 3rd dose of ETX2514 and sulbactam will be administered on Day 2 .
Mean clearance (CL) in blood | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analysis predose, and 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third (last) dose.
Ratio of AUC 0-6 for ELF to the corresponding AUC0-6 Plasma | Predose, 1,2,2,5, 2.95, 3.05, 3.25, 3.5, 4, 5, and 6 hours after the start of the third dose (last dose) on Day 2
  defined as the area under the concentration versus time curve from time zero to 6 hours. Venous blood will be collected for ETX2514SUL pharmacokinetic (PK) analysis predose and after the 3 dose. The 3rd dose of ETX2514 and sulbactam will be administered on Day 2. Bronchoalveolar lavage fluid will be collected for ETX2514SUL PK at 1, 2.5, 3.25, 4, or 6 hours after the 3 dose (last dose) on Day 2.

SECONDARY OUTCOMES:
Number of participants with any non serious adverse event (AE) | Day 1-14
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Number of participants with any serious adverse event (SAE) | Day 1- 14
  An SAE is defined as any event that results in death; is immediately life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Change from Baseline in electrocardiogram (ECG) parameters at the indicated time points | Day 1, 2, and 4
  Change in baseline is calculated as the post-baseline value minus the baseline value
Change from baseline in vital signs at the indicated time points | Days 1, 2,and 4
  change from baseline in calculated as the post baseline value minus the Baseline value
Number of participants with abnormal, clinical significant hematology and chemistry laboratory values at the indicated time points | Day 1-14
  Change from baseline is calculated as the post-Baseline value minus the Baseline value

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates, PA, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodvold KA, Gotfried MH, Isaacs RD, O'Donnell JP, Stone E. Plasma and Intrapulmonary Concentrations of ETX2514 and Sulbactam following Intravenous Administration of ETX2514SUL to Healthy Adult Subjects. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e01089-18. doi: 10.1128/AAC.01089-18. Print 2018 Nov. PMID 30126953